CLINICAL TRIAL: NCT07110467
Title: Nursing Intervention of Blinking Exercises as a Non-Pharmacological Approach to Alleviate Dry Eye and Enhance Daily Life in Older Adults: A Quasi-Experimental Study
Brief Title: Nursing Intervention of Blinking Exercises to Alleviate Dry Eye and Enhance Daily Life in Older Adults
Acronym: blinking dry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norther Private Collage of Nursing (Other)
Responsible Party: Principal Investigator, Amal, Associate professor, Norther Private Collage of Nursing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID/Zu.Nur.REC #: 272
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Daily Activities; Eye Health

STUDY DESIGN:
Intervention Model Description: the participants divided into two group experimental and placebo group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blinking excelsis group (Experimental): The study group were divided into small training groups with 3-5 older adult for each group. Two sessions were needed for each group each session took about 1- 2hrs.
  • The 1st session included (definition, causes, signs & symptoms, risk factors, complications, prevention, and management of eye dryness and the 2nd session covered the recommended exercises for reducing eye dryness including (Eye gaze exercise, Right and left eye movement exercise, eye rise and fall exercise, eye-crossing exercise, eye control exercise, eye pressure exercise, eye rotation exercise, and eye relaxation exercise).
  This group was instructed to instill artificial tears and perform blinking exercises three- five times a day for 4 weeks.
  Interventions: Procedure: blinking exercises
- control group (Sham Comparator): this group receive moisturizing eye drop only
  Interventions: Procedure: blinking exercises

INTERVENTIONS:
Procedure: blinking exercises — The study group was instructed to instill artificial tears and perform blinking exercises three- five times a day for 4 weeks.

SUMMARY:
The study aimed to evaluate the effect of blinking exercises in improving eye dryness and daily life in older adults. Participants aged 60 years and older of both genders, diagnosed with dry eyes and patients who were alert and able to communicate.

DETAILED DESCRIPTION:
The Research hypotheses include H0: Nursing interventions of blinking exercise do not affect the level of dry eyes and daily life in older adults.

H1: Nursing interventions of blinking exercise affect the level of dry eyes and daily life in older adults.

Participants were divided into two groups (study and control). Both groups were asked to fill out all questionnaires before and after the study using the same tools. In the control group, older adult receives routine care, which was provided by the hospital as examination, application of moisturizing eye drops three- five times Aday for 4 weeks . Participants were asked to answer a post-test using the same pre-test questionnaires. And the study group were divided into small training groups with 3-5 older adult for each group. Two sessions were needed for each group each session took about 1- 2hrs.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and older of both genders, diagnosed with dry eyes and patients who were alert and able to communicate.

Exclusion Criteria:

* Patients underwent refractive surgery procedures.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
change in quality of life | 4 weeks following the end of treatment
  Impact Dry Eye Everyday Life Questionnaire it include 3 domains (daily activity limitations, emotional wellbeing, and work limitations), a scale score is calculated between 0 (representing total impairment) and 100 (representing no impairment). The daily activities sub-domain is the quality of life instrument. It is comprised of 27 items, each item had five answers "strongly agree" is scored as 1, "agree" is scored as 2, "neutral" is scored as 3, "disagree" is scored as 4, and "strongly disagree" is scored as 5. The greater score indicate high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Assistance professor, phd, Study Director — Cairo University
Locations (1):
- Norther Private Colleague of Nursing, Arar, Norther Border, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Analysis of influencing factors of dry eyes after cataract surgery and construction of a prediction model — https://pmc.ncbi.nlm.nih.gov/articles/PMC11558407/